CLINICAL TRIAL: NCT00173056
Title: The Factors Predicting Change of Peritoneal Transport Characters in Peritoneal Dialysate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700731
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2004-12

CONDITIONS: Peritoneal Fibrosis
Keywords: Peritoneal dialysis
MeSH Terms: conditions — Peritoneal Fibrosis

SUMMARY:
Peritoneal fibrosis (PF) is one of the most serious complications after long-term continuous ambulatory peritoneal dialysis (CAPD). Human peritoneal fibroblast (HPFB) and extracellular matrix (ECM) deposition is the most possible causes leading to PF. ECM are mainly synthesized from HPFB and human peritoneal mesothelial cells (HPMC). In the PF process, there is decrement in the quantity of HPMC, loss of permeability for lower molecules, and eventually ultrafiltration failure. This phenomena will result in technique failure.

High glucose content of the dialysate and peritonitis have been claimed as major stimulants to the development of PF. In each episode of peritonitis, the number of HPMC will decrease. On the other hand, ECM production will be reinforced by the inflammatory cytokines secreted by the white cells or HPMC per se. High glucose dialysate will induce the above process with more chronic stimulation, and PF followed by technique failure is inevitable.

Peritoneal fibrosis is definitively diagnosed with peritoneal biopsy, but this is inconvenient for most patients. Besides, pathology changes will be noted only after a substantial loss of peritoneal function. The peritoneal equilibration test (PET) is usually used as the index of peritoneal function. However, in the chronic process, PET change is also slow and is unable to be a parameter for treatment outcome. In this study, the factors predicting PET change will be searched, and they could be an index for evaluation and even a marker of preventing or treating PF.

In this project, peritoneal dialysis (PD) dialysate will be collected during an annual PET in each PD patient in the National Taiwan University Hospital (NTUH). Some cytokines that will be measured include vasculoendothelial growth factor, hyaluronan, transforming growth factor-β, procollagen, and cancer antigen-125. The same test and measurement will be performed during PET in the next year. The factors which affect PET results will be analyzed such as cytokines, glucose exposure, peritonitis incidence, PD duration, gender, age. The investigators will try to find a convenient acute reactive marker for preventing or treating PF to monitor the PET change clinically.

ELIGIBILITY:
Inclusion Criteria:

* All PD patients

Exclusion Criteria:

* Peritonitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jenq-Wen Huang, MD, Principal Investigator — Department of Internal Medicine, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan